CLINICAL TRIAL: NCT03704649
Title: Evaluating the Effectiveness of a Participatory Video Nutrition Education Trial on Nutrition Literacy With Adolescent Girls in the Upper Manya Krobo District, Ghana.
Brief Title: Evaluating a Participatory Nutrition Education Model on Nutrition Literacy of Adolescent Girls in Rural Ghana.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: University of Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QES01
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition; Adolescent Development; Adolescent Behavior
Keywords: Nutrition; Literacy; Education; Adolescent; Girl; Participatory; Video; Ghana
MeSH Terms: conditions — Malnutrition; Adolescent Behavior; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard nutrition education (No Intervention): The comparison group for the participatory video intervention.
- Participatory nutrition education (Experimental): Intervention arm integrates participatory video model to standard girls' club sessions to promote nutrition education.
  Interventions: Behavioral: Participatory video

INTERVENTIONS:
Behavioral: Participatory video — Participatory video education is an intervention model that gives communities the film-making skills necessary to make videos that can be used in nutrition promotion. For the purposes of this study, we will be using a participatory video model as an approach to educate participants in a school-based girls club on nutrition education topics. Participants are taught how to use film equipment and accompanied to draft scripts, create characters, video-record the shots, and act (if they wish) in the video. These videos will be used in the group as a means of sharing nutrition information with students and in stimulating discussion around the nutrition topic.
  Other Names: Community-led video education
  Arms: Participatory nutrition education

SUMMARY:
Adolescent girls in the Upper Manya Krobo (UMK) district, Ghana are disproportionately burdened by ill-health in relation to their male counterparts. Research also shows that this demographic lacks access to nutrition education and health services. This research aims to assess the feasibility and influence of an intervention that utilizes a participatory video education model on adolescent girls' nutrition knowledge, dietary habits and health behaviour. To address our research objectives, we will conduct a school-based cluster randomized control pilot trial with adolescent girls, 12-16 years of age, who are part of existing girls' clubs in 20 schools of the Upper Manya Krobo district. The intervention group (10 schools) will use a participatory video education model and the control group consists of standard-of-care education received in regular girls' club gatherings. The intervention groups develop a storyboard and produce a short 5-7 minute film on a nutritional issue. These videos can be used by teachers as a means of sharing nutrition information with students and in stimulating discussion around the nutrition topic. Baseline and end line surveys will be conducted to assess nutrition literacy indicators and nutrition behaviour. We will use surveys to assess nutritional knowledge and attitude; food frequency questionnaire to record dietary intakes; and in-depth interviews with participants and school staff to assess challenges and strengths of the nutrition education model being delivered.

DETAILED DESCRIPTION:
Although there are a number of health and nutrition services targeted to adolescent girls in rural Ghana, there continues to be a high prevalence of anemia, preventable ailments, and teen pregnancies among adolescent girls in the Upper Manya Krobo district. This project builds on a health literacy framework and social cognitive theory and explores salient features in nutrition education delivery with adolescent girls in the Upper Manya Krobo district of Ghana, and investigates their influence on nutritional knowledge and behaviour.

The primary research objective is (1) to assess the feasibility of a participatory nutrition education model in the Upper Manya Krobo district and, (2) to determine if there is a difference in adolescent girls' nutrition literacy between the intervention and control groups. The research will provide a process evaluation and offer insight into a replicable and feasible protocol that can implemented in other schools. We hypothesize that there will be a difference in nutrition literacy indicators and dietary patterns between intervention and control groups.

To address our research objectives, we will conduct a school-based cluster randomized control pilot trial with adolescent girls, 12-16 years of age, who are part of existing girls' clubs in 20 schools of the Upper Manya Krobo district. Eligible clusters consist of primary and/or junior high schools in UMK district that are implementing standardized girls' clubs and who intend to continue to implement girls' clubs for the upcoming 2018-2019 school year (n = 59). Clusters will be stratified based on 1) the presence of the school feeding program and 2) accessibility to the school. Accessibility will be based on the quality of roads and time needed to travel to the cluster from the district capital, Asesewa. After stratification, clusters will be randomized into control and treatment arms. In each cluster, approximately 20 female adolescent girls' club participants who are 12-16 years of age will be randomly selected and enrolled in the study through seeking informed guardian's consent and adolescent's assent.

The control groups (10 schools) represent the standard-of-care. Participants in these clubs meet on a weekly basis during designated time for club activities in the school schedule. With the guidance of their club facilitator they talk about a variety of health and nutrition topics. The intervention groups (10 schools) will follow a similar curriculum and will include a participatory video education model. The intervention groups develop a storyboard and produce a short 5-7 minute film on a nutritional issue where they are the individuals who draft the script, create the characters, video-record the shots, and act (if they wish) in the video. These videos will be used in the group as a means of sharing nutrition information with students and in stimulating discussion around the nutrition topic.

Data Collection Procedures

Phase 1: Baseline survey and weight/height.

Baseline surveys will be conducted to assess nutrition literacy indicators and nutrition behaviour. Survey questionnaires will be administered at baseline by trained research assistants using electronic tablets. The Open Data Kit (ODK) software will be downloaded onto Samsung Tab3 tablets that will be used to record survey questionnaire responses. This survey will take about 30-45 minutes and will be conducted in a private location on the student's school campus. We will use surveys to assess nutritional knowledge and attitude; questionnaires to record dietary intakes. She will be asked about herself and her family (for example, age, schooling, occupation), what she knows about food and nutrition, her diet, and how she spends her free time. Her weight and height will be taken.

Phase 2: Intervention.

The proposed intervention entails the active engagement of key community members, community-based organizations and governmental institutions in the UMK district. A community advisory board (CAB) is formed by key stakeholders, including health professionals, community health workers, government officials, and influential community members. Their primary role is to follow the development of the project, help to identify key health and nutrition messages, to ensure the credibility of the health message being disseminated, and to help strengthen community connections necessary for the seamless execution of the research-related activities.

A minimum of two girl club facilitators per school will attend a training to review health and nutrition themes dictated in the girls' club standard curriculum. Facilitators from intervention schools will participate in additional film production workshops where they are trained on how to write storyboards and scripts, and use microphones and cameras to make short 5-7 minute films. In the intervention girls' clubs sessions, the facilitators lead a discussion on nutrition topics and assist the girls to develop a scenario, storyboard and script for the educational video they will produce. A script is written in the local Krobo dialect and auditions are held in their club to cast the various roles. After the video is produced, it is viewed and approved by members of the CAB, to ensure that material is culturally appropriate and that the nutrition information is accurate. The video is made available to girls' club teachers who will screen it for the students with the use of a battery operated pico projector and speakers, after which the audience is prompted to reflect on the video being watched. Each intervention group will produce two videos on the nutrition topics covered in the girls' club session.

Throughout this time, observations will be gathered regarding attendance and the content of the nutrition messages delivered in the girls' club sessions.

Phase 3 - In-depth interview and Focus group discussion.

In-depth interviews will be conducted with participants. Whether the female participant is in the intervention group or not, she may be selected to be interviewed based on the recommendation of her club facilitator through purposive typical case sampling. This is done so as to gain insight on the influence of the educational curriculum and/or intervention on the average student. The purpose of this interview is to better understand her experience in the girls' club, what nutrition information she remembers from the lessons, what helped her and what challenges she faced in putting into practice what she learned. The most significant change methodology is used in the interview guide design. The interview will be about 30 minutes.These interviews will be conducted in a private location at their schools after the guardian's informed consent and participant informed assent is given.

Focus group discussions will also be conducted with staff and community members that were associated to the girls' club activities. The purpose of this focus group discussion is to better understand their experience with the girls' club sessions. Focus group discussions will provide insights into helpful aspects or challenges that were faced when supporting the girls' club activities. Other questions will focus on the changes they may have noticed in the participant's understanding and attitude towards nutrition and changes in their eating behaviour. The focus group discussion will be about 30-45 minutes.

Phase 4 - Post-intervention surveys and weight/height.

Surveys will be conducted with the girl participants at the end of the school year when the intervention is completed. Surveys will be used to assess changes in nutrition literacy indicators and nutrition behaviour.

Data management and analysis.

Data from these surveys will be downloaded into a password protected and secured laptop at the end of every day and then deleted off the tablet. Data will be backed up on an external hard drive that is located in a locked cabinet of the offices in the Nutrition Research and Training Centre in Asesewa.

Each participant will be given a code number to protect the participant's identity. With their guardian's consent and the participant's assent interviews will be audio-recorded and then translated and written out for our records. Audio files of interviews will be deleted off equipment after the study is finished and they are only for the use of the researcher. All equipment used in collecting or storing data will be password protected. Hard copies of consent forms, transcripts, and demographic data will be stored in a locked storage cabinet at University of Ghana and McGill University. In addition to the researchers, community health workers and school teachers tied to the girls' clubs will have a copy of the final films made by the girls to use in their educational activities.

ELIGIBILITY:
Inclusion Criteria:

* Is a female participant of girls' club in the school that was randomly selected to participate in the study
* Resides in the Upper Manya Krobo district.
* Is 12 to 16 years of age

Exclusion Criteria:

* Does not speak local dialect - Krobo.

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 351 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change in nutrition literacy indicators | 8-10 months
  Survey questionnaire will record functional, interactive and critical nutrition literacy indicators that will be used to assess change in nutrition literacy outcome.

SECONDARY OUTCOMES:
Change in psychological health behaviour change indicators | 8-10 months
  Survey questionnaire will record psychological health behaviour change indicators such as changes in self-efficacy and intention to change behavior.
Change in dietary choices | 8-10 months
  Survey questionnaire will record changes in dietary habits through the use do a food frequency questionnaire.
Feasibility - process evaluation | 8-10 months
  Input into the feasibility of the protocol emerging from focus group discussions and in-depth interviews with staff and participants

CONTACTS AND LOCATIONS:
Overall Officials: Grace Marquis, PhD, Principal Investigator — McGill University
Locations (2):
- McGill University, Montreal, Quebec, Canada
- University of Ghana, Legon, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghadirian MZ, Marquis GS, Dodoo ND, Andersson N. Ghanaian Female Adolescents Perceived Changes in Nutritional Behaviors and Social Environment After Creating Participatory Videos: A Most Significant Change Evaluation. Curr Dev Nutr. 2022 Jun 16;6(8):nzac103. doi: 10.1093/cdn/nzac103. eCollection 2022 Aug. PMID 36060219